# MODIFICAZIONI ENDOMETRIALI NELLE PAZIENTI CON CARCINOMA DELLA MAMMELLA

# **CENTRO PROPONENTE/SPONSOR dello studio (no-profit):**

# IFO-Istituti Fisioterapici Ospitalieri Roma

Via Elio Chianesi, 53 – 00144 ROMA

# PRINCIPAL INVESTIGATOR (P.I.):

Dr. Benito Chiofalo

UOC Ginecologia IRE – <u>Direttore Dr. E. Vizza</u>

Tel: 06-52666970

mail: benito.chiofalo@ifo.it

#### **PARTECIPANTI IFO**

Dr. Mario Russo

UOC Ginecologia IRE (specializzando Federico II di Napoli)

Email: mariorussom39@gmail.com

# Elaborazione statistica e Monitoraggio Supporto Studi Clinici:

Dr.ssa Francesca Sperati Email: francesca.sperati@ifo.it Dr.ssa Federica Falcioni Tel. 06-5266.5353

#### **PAGINA FIRME**

Dichiaro di aver letto il protocollo in oggetto ed accetto di condurre lo studio secondo quanto riportato, secondo i principi etici per la conduzione della Sperimentazione Medica in Soggetti Umani adottati nella Dichiarazione di Helsinki, ICH-GCP, nonché conformemente alla normativa vigente in materia di studi clinici e di trattamento dati personali.

Accetto di condurre lo studio in prima persona e/o di supervisionarlo.

Firma PI/Sperimentatore:

Inoltre garantisco che tutti coloro che mi assisteranno nella conduzione dello studio avranno accesso al protocollo dello studio ed eventuali emendamenti, a tutte le informazioni e documenti secondo quanto pertinente, e saranno consapevoli delle loro responsabilità.

| PI CENTRO PROMOTORE: | |
|---|---|
| Ospedale/Istituto: IFO-IRE Istituto Nazionale Tumori Regina Elena PI/Sperimentatore: | _ |
| Firma PI/Sperimentatore: Data: | l |
| CENTRO DI RIFERIMENTO/PI locale: Dichiaro di aver letto il protocollo in oggetto ed accetto di condurre lo studio secondo quanto riportato secondo i principi etici per la conduzione della Sperimentazione Medica in Soggetti Umani adottati nelli Dichiarazione di Helsinki, ICH-GCP, nonché conformemente alla normativa vigente in materia di studi clinice e di trattamento dati personali. Accetto di condurre lo studio in prima persona e/o di supervisionarlo. Inoltre garantisco che tutti coloro che mi assisteranno nella conduzione dello studio avranno accesso a protocollo dello studio, ad eventuali emendamenti, a tutta la relativa documentazione pertinente, e sarann consapevoli delle loro responsabilità. | a<br>ci |
| Ospedale/Istituto: | |

Data: |\_\_\_\_|

# Introduzione/Razionale (introduzione al problema anemia)

Il carcinoma mammario rappresenta un fattore di rischio per le patologie endometriali [1]. Non sono ben noti i fattori che determinano la gran parte delle patologie endometriali, ma è noto che esistono dei fattori di rischio comune tra la patologia mammaria e quella endometriale, sia costituzionali, ma specialmente ormonali (iperestrogenismo). Infatti l'ambiente iperestrogenico rappresenta anche il target principale delle terapie ormonali nel carcinoma della mammella ormonosensibile [2]. Selective estrogen receptor modulators (SERMs) e inibitori dell'aromatasi (Als) mirano a ridurre l'azione degli estrogeni a livello mammario, ma poco si conosce sull'effetto di questi farmaci sugli altri tessuti bersaglio.

Le modificazioni endometriali indotte dal tamoxifene sono un'ipertrofia dello stroma, modificazioni cistiche dell'endometrio, molto caratteristiche, osservabili in quasi tutte le pazienti che si sottopongono a questa terapia.

Queste modificazioni sono benigne, alcuni autori suggeriscono che il tamoxifene aumenti l'incidenza di altre patologie endometriali uterine benigne [3-5] e di carcinoma dell'endometrio [6].

Due precedenti studi retrospettivi condotti su tre diversi gruppi di pazienti con carcinoma mammario sottoposte a terapia con Als, con tamoxifene o a nessuna terapia ormonale, hanno evidenziato come non ci sia un aumento dell'incidenza di carcinoma dell'endometrio nelle pazienti che assumono tamoxifene rispetto agli altri gruppi [7].

Non esistono in letteratura studi clinici prospettici, che abbiano valutato i suddetti aspetti.

# Scopo dello Studio e Razionale Scientifico

L'obiettivo dello studio è di valutare l'incidenza di carcinoma dell'endometrio in tre diversi gruppi di pazienti con carcinoma mammario.

Ulteriore obiettivo dello studio è quello di identificare fattori di rischio ecografici, altamente indicativi di carcinoma dell'endometrio.

# Disegno dello studio

Studio osservazionale prospettico di coorte, multicentrico.

Arruoleremo tutte le pazienti con storia personale positiva di carcinoma mammario che afferiscono agli ambulatori di ginecologia dei centri partecipanti e che risponderanno ai requisiti previsti.

## Obiettivi dello studio

## Obiettivo principale:

L'obiettivo dello studio è valutare l'incidenza di carcinoma dell'endometrio in pazienti con storia di carcinoma mammario in tre diversi gruppi di pazienti con carcinoma mammario (SERMs users, Als users e pazienti che non fanno uso di terapia ormonale (NT))

## Obiettivi secondari:

Ulteriore obiettivo dello studio è quello di identificare fattori di rischio ecografici e isteroscopici, altamente indicativi di carcinoma dell'endometrio.

# Popolazione in studio:

#### Criteri di inclusione:

- Età > 18 anni
- Pazienti con storia personale positiva di carcinoma della mammella che afferiscono agli ambulatori di ginecologia dei centri partecipanti per visite ginecologiche
- consenso informato scritto

#### Criteri di esclusione:

- Pazienti con storia personale di altri tumori ormono-sensibili.
- Pazienti portatrici di dispositivo intrauterino.
- Pazienti che hanno eseguito ormono-terapia (diversa da quella oggetto di studio) nei 5 anni precedenti.
- Pazienti con anamnesi positiva per tecniche di procreazione medicalmente assistita.
- Pazienti con sindrome di Lynch, mutazioni patogenetiche del gene BRCA e altre sindromi eredofamiliari ad aumentato rischio oncologico.

# Metodi e Procedure

Tutte le pazienti arruolate verranno sottoposte, secondo la corretta pratica clinica, a ecografia transvaginale e visita ginecologica con cadenza annuale. Se a seguito dell'esame ecografico verrà evidenziata una sospetta patologia endometriale o uno spessore endometriale aumentato ( > o uguale a 10mm se TAM user, oppure > o uguale a 4 mm se non TAM user), oppure, sintomatiche per perdite ematiche atipiche dai genitali esterni (spotting, menometrorragie non disfunzionali, perdite ematiche vaginali in post-menopausa) con ecografia transvaginale negativa, verranno sottoposte ad isteroscopia diagnostica (office o sala operatoria)[8].

La descrizione di ogni procedura verrà attentamente analizzata.

Le pazienti verranno quindi suddivise in tre gruppi sulla base dei criteri clinici ed ecografici descritti.

**Gruppo 1**: Pazienti con carcinoma della mammella SERMs user

Gruppo 2: Pazienti con carcinoma della mammella Als user

**Gruppo 3**: Pazienti con carcinoma della mammella che non fanno uso di terapia ormonale (NT)

I dati relativi ai risultati anatomo patologici delle biopsie endometriali eseguite verranno analizzati al fine di valutarne l'incidenza di carcinoma endometriale e/o iperplasia endometriale atipica nelle pazienti partecipanti allo studio.

Per ogni paziente saranno quindi raccolte ed elaborate le seguenti principali categorie di dati:

dati anagrafici e socio-demografici (quali età/anno di nascita)

dati clinici/sanitari (anamnesi remota e prossima, anamnesi ostetrica)

dati anatomo-patologici (quali diagnosi, stadio, ecc)

dati relativi ad eventuali trattamenti (tipo di trattamento, periodo, ecc)

dati relativi alle valutazioni ed esami effettuati (in particolari esame obiettivo, ecografia transvaginale, eventuale isteroscopia)

I dati raccolti saranno opportunamente codificati ed inseriti in un apposito database, la cui configurazione sarà sotto la responsabilità del Centro Proponente.

#### **DIMENSIONE DEL CAMPIONE E METODI STATISTICI**

# Calcolo numerosità campionaria

Per determinare la numerosità campionaria necessaria abbiamo basato le nostre stime sull'incidenza di cancro dell'endometrio.

Lo studio prevede il confronto tra tre gruppi di pazienti: un gruppo di controllo (nessun trattamento (NT)) e due gruppi trattati (con TAM e AI, rispettivamente). Il numero totale dei confronti di interesse è pari a tre. Per ogni gruppo abbiamo ipotizzato i seguenti valori di incidenza del cancro dell'endometrio, partendo da uno studio retrospettivo [7]:

NT group: 11.1%;TAM group: 3.8%;Al group: 0.1%.

Abbiamo quindi fissato i valori dei seguenti parametri:

- una potenza statistica (1-β) pari all' 80%
- un livello di significatività  $\alpha$  pari a 0.05 aggiustata secondo la correzione di Bonferroni (=  $\alpha$  / #confronti) per confronti multipli:in questo caso 0.05 / 3 = 0.017

Utilizzando il test a due code di Fisher, il numero stimato di pazienti per ogni confronto sarà il seguente:

| Confronto di interesse | N1 | N2 |
|------------------------|-----|-----|
| NT vs TAM | 281 | 281 |
| NT vs Al | 84 | 84 |
| TAM vs Al | 267 | 267 |

Pertanto il numero totale di pazienti da arruolare sarà 829 (281 pe i gruppi NT e TAM e 267 per il gruppo AI).

# Analisi statistiche

Calcoleremo le statistiche descrittive per tutte le variabili di interesse: in particolare, riporteremo le variabili continue con le loro medie e deviazioni standard (±SD) e le variabili categoriche con frequenze assolute, relative e percentuali. Eseguiremo il test di normalità di Kolmogorov-Smirnov per tutte le variabili continue. Per confrontare le variabili, utilizzeremo i test più adatti in base alla natura della distribuzione dei dati. Useremo un modello di regressione logistica univariata per identificare le variabili che potrebbero avere un ruolo nel rischio di sviluppare il cancro dell'endometrio. Verrà utilizzato un modello di regressione logistica multivariata con variabili predittive che saranno significative nelle analisi univariate. L'analisi di sopravvivenza sarà eseguita utilizzando il metodo di Kaplan-Meier e il modello di regressione dei rischi proporzionali di Cox. Tutte le analisi statistiche saranno eseguite con l'ausilio del software statistico SPSS versione 21 (SPSS inc., Chicago IL, USA). Un p-value <0.05 sarà considerato statisticamente significativo.

# Risultati attesi, loro potenziale significato e spendibilità clinico-scientifica

Ridurre il tasso di esami isteroscopici e di biopsie endometriali superflui nelle pazienti con pregresso carcinoma della mammella. Individuare marcatori ecografici (cut-off endometriale) indicativi di

patologie endometriali nelle pazienti con carcinoma della mammella. Orientare in maniera evidence-based il percorso diagnostico ginecologico nelle pazienti con pregresso carcinoma della mammella.

## **DURATA** prevista

Periodo di arruolamento: 1 anno

Follow-up/raccolta dati: almeno 3 mesi dall'arruolamento

Durata totale: 1,5 anni

#### **ASPETTI ETICI E AMMINISTRATIVI**

La conduzione dello studio avverrà in accordo con i principi della Buona Pratica Clinica ("Good Clinical Practice"), nonché secondo quanto richiesto dalle autorità regolatorie e dalle principali normative europee e nazionali applicabili.

E' responsabilità del PI dello studio garantire che lo stesso sia condotto in accordo alla Dichiarazione di Helsinki, alle GCP, ed alla normativa vigente al riguardo; nonché il rispetto della normazione in tema di tutela della persona di cui si trattano i dati personali secondo il Regolamento UE 2016/679 e Codice Privacy domestico.

Prima di essere attivato, lo studio dovrà essere sottoposto al Comitato Etico di riferimento del centro coordinatore/locale per opportuno parere, nonché dell'eventuale autorizzazione amministrativa (se pertinente).

#### **Emendamenti**

Nessun cambiamento al protocollo può essere effettuato senza averlo preventivamente sottoposto al Comitato del centro coordinatore (e locale/di riferimento) per opportuno parere e/o presa d'atto.

#### **Data Quality Assurance**

Il promotore è responsabile dell'implementazione e del mantenimento dei sistemi di controllo di qualità per garantire che lo studio sia condotto e che i dati siano generati, documentati (registrati) e riportati in conformità con il protocollo, con le GCP ed i requisiti normativi applicabili. Il promotore potrà eseguire un monitoraggio per verificare la conduzione dello studio, compreso un monitoraggio dei dati per verificare l'aderenza al protocollo e la correttezza delle informazioni raccolte.

# Consenso informato

Il ricercatore responsabile dello studio e/o un Suo delegato dovrà ottenere il consenso informato (ICF) scritto da parte delle partecipanti (e/o dalla persona che acconsente a nome del soggetto) prima di attivare qualsiasi procedura ad esso relativa.

Tutti gli ICF firmati (e compilati in ogni parte secondo quanto opportuno), devono essere conservati tra la documentazione dello studio presso ogni centro secondo le modalità e le tempistiche previste dalla normativa e dalle disposizioni vigenti in materia.

Il modulo di consenso originale firmato e datato dal soggetto interessato e/o dalla persona che acconsente a nome del soggetto deve essere conservato nei fascicoli di studio dello sperimentatore presso il centro di riferimento.

La documentazione che il processo di consenso informato e la sottoscrizione della relativa dichiarazione consenso informato è avvenuto prima dell'ingresso della paziente nello studio e dell'attivazione di qualsiasi procedura ad esso relativa deve essere registrata nei documenti di origine del soggetto.

## Revoca consenso

I soggetti interessati hanno il diritto di revocare il consenso alla partecipazione allo studio rilasciato in ogni momento e per qualsiasi motivo.

In tal caso non saranno raccolti ulteriori dati relativi alle partecipanti, fermo restando l'utilizzo di quelli precedentemente raccolti al fine di non pregiudicare i risultati della ricerca; la revoca del consenso alla

partecipazione allo studio non pregiudica infatti la liceità del trattamento svolto sulla base del consenso precedentemente prestato e avrà come unico effetto la cessazione del trattamento dei dati personali dell'interessato per il futuro.

## Confidenzialità dei dati

Il personale coinvolto nella conduzione del presente studio garantirà il rispetto della confidenzialità dei dati di tutti le pazienti incluse/arruolate.

Saranno seguite le regole dettate dal Regolamento Europeo 2016/679, noto come GDPR (General Data Protection Regulation) e dal Codice Privacy e ss.mm.ii. per la protezione degli individui in relazione alla gestione dei dati personali ed alla libera circolazione degli stessi. Gli sperimentatori dovranno garantire che sia mantenuto il rispetto della riservatezza delle pazienti. Sulle CRF e sugli altri documenti la paziente sarà identificata mediante un codice univoco.

In accordo con quanto prescritto dalla legislazione italiana e dalle linee guida ICH/GCP, gli sperimentatori consentiranno a rappresentanti delle agenzie regolatorie e del Comitato Etico, del Promotore e/o agli addetti al monitoraggio opportunamente autorizzati, accesso diretto per la revisione della documentazione originale delle pazienti, per verificare il rispetto delle procedure e la veridicità dei dati.

## Raccolta e gestione dati

Ad ogni paziente sarà assegnato un codice identificativo le cui modalità saranno definite dal promotore/PI principale dello studio; solo il ricercatore responsabile dello studio presso il centro ed i suoi collaboratori, nonché il personale e/o addetti al monitoraggio/verifiche opportunamente autorizzati, saranno in grado di risalire all'identità dei soggetti arruolati/reclutati.

Saranno adottate tecniche di cifratura/codici identificativi o di pseudonimizzazione che non renderanno direttamente riconducibili i dati ai soggetti interessati, permettendo di identificare questi ultimi solo in caso di necessità

I dati (comprese le immagini radiologiche) saranno raccolti, conservati, utilizzati, trattati da parte del personale autorizzato nonché trasmessi al promotore/coordinatore e/o coloro che collaborano nello svolgimento dello studio, secondo le modalità e le tempistiche vigenti e definite al riguardo, garantendone la qualità, l'integrità, la sicurezza, la disponibilità e la tracciabilità, sotto la responsabilità del PI locale, facendo in modo che venga sempre assicurato il rispetto e la conformità con quanto richiesto dalla normativa per il trattamento dei dati personali e/o da tutta la normativa di riferimento vigente.

È responsabilità del ricercatore/PI locale dello studio far sì che i dati siano raccolti in modo appropriato e completo.

L'accesso ai sistemi informatici ed ai locali ove essi sono custoditi/trattati sarà controllato mediante idonee misure di sicurezza e possibile solo al personale autorizzato ed opportunamente identificato.

Tutte le informazioni raccolte, così come i risultati delle analisi condotte, saranno trattate/trattati con la massima riservatezza.

Il Promotore/centro adotterà opportune misure tecniche ed organizzative per garantire un livello adeguato di sicurezza dei dati trattati nell'ambito dello studio, nonché specifiche misure ed accorgimenti tecnici per incrementare lo stesso e per prevenire la diffusione dei dati personali o il loro utilizzo da parte di soggetti non autorizzati.

I dati, il materiale e la documentazione relativa allo studio saranno conservati da parte del Promotore/centro, ognuno secondo propria competenza, per il periodo di tempo necessario per conseguire le finalità dello studio conformemente a quanto stabilito dalla normativa e dai regolamenti che disciplinano la materia (per un periodo di 5 anni dalla conclusione dello studio o per un periodo più lungo, secondo quanto stabilito dalle leggi e/o dai regolamenti applicabili) e/o per eventuale riuso per finalità di ricerca scientifica, conformemente a quanto stabilito dalla normativa e dai regolamenti che disciplinano la materia, secondo modalità tali da garantirne comunque la riservatezza e la sicurezza delle informazioni contenute.

Al termine del periodo di conservazione i dati personali saranno cancellati/anonimizzati, a condizione che non sussistano ulteriori obblighi di legge; potranno essere conservati per periodi più lunghi esclusivamente a fini di archiviazione nel pubblico interesse, di ricerca scientifica o storica o a fini statistici, fatta salva l'attuazione di misure tecniche e organizzative adeguate richieste dal GDPR/della normativa applicabile a tutela dei diritti e delle libertà del soggetto interessato.

Il Titolare potrà conservare i dati illimitatamente ma unicamente previo processo di anonimizzazione che non consenta in alcun modo di rendere identificato o identificabile ogni singolo arruolato/interessato. Infine, ad ogni Titolare dello studio spetteranno tutti e ciascuno gli adempimenti nascenti dalla normazione europea ed italiana in tema di tutela dei dati personali, ivi inclusi i provvedimenti del Garante per la protezione dei dati personali.

#### Proprietà dei dati

Il Promotore è proprietario esclusivo di tutti i dati e le informazioni derivanti dallo studio, inclusi risultati, scoperte, know-how e simili.

# Uso e pubblicazione dati

I risultati principali dello studio saranno pubblicati su riviste nazionali e/o internazionali e potranno essere presentati in convegni scientifici, studi statistici, pubblicazioni scientifiche, in tabelle e grafici, ecc. in forma aggregata ed anonima, riferiti a gruppi di persone e mai a singoli individui.

Ad ogni centro partecipante sarà garantita visibilità proporzionale alla effettiva partecipazione.

# Bibliografia

- 1. Le Donne M, Lentini M, De Meo L, Benedetto V, Mesiti M. Uterine pathologies in patients undergoing tamoxifen therapy for breast cancer: ultrasonographic, hysteroscopic and histological findings. Eur J Gynaecol Oncol. 2005;26:623–626.
- 2. Jordan VC, Assikis VJ. Endometrial carcinoma and tamoxifen: clearing up a controversy. Clin Cancer Res. 1995;1:467–472.
- 3. Dallenbach-Hellweg G, Hahn U. Mucinous and clear cell adenocarcinomas of the endometrium in patients receiving antiestrogens (tamoxifen) and gestagens. Int J Gynecol Pathol. 1995;14:7–15.
- 4. Fung MF, Reid A, Faught W, et al. Prospective longitudinal study of ultrasound screening for endometrial abnormalities in women with breast cancer receiving tamoxifen. Gynecol Oncol. 2003;91:154–159.
- 5. Liedman R, Lindahl B, Andolf E, Willen R, Ingvar C, Ranstam J. Disaccordance between estimation of endometrial thickness as measured by transvaginal ultrasound compared with hysteroscopy and directed biopsy in breast cancer patients
- 6. Cohen I, Altaras MM, Shapira J, et al. Time-dependent effect of tamoxifen therapy on endometrial pathology in asymptomatic postmenopausal breast cancer patients. Int J Gynecol Pathol. 1996;15:152–157.
- 7. LE Donne M, Alibrandi A, Ciancimino L, Azzerboni A, Chiofalo B, Triolo O. Endometrial pathology in breast cancer patients: Effect of different treatments on ultrasonographic, hysteroscopic and histological findings. Oncol Lett. 2013 Apr;5(4):1305-1310. doi: 10.3892/ol.2013.1156. Epub 2013 Jan 28. PMID: 23599784; PMCID: PMC3629067.
- 8. Saccardi C, Gizzo S, Patrelli TS, Ancona E, Anis O, Di Gangi S, Vacilotto A, D'Antona D, Nardelli GB. Endometrial surveillance in tamoxifen users: role, timing and accuracy of hysteroscopic investigation: observational longitudinal cohort study. Endocr Relat Cancer. 2013 Jun 24;20(4):455-62. doi: 10.1530/ERC-13-0020. PMID: 23629476.